CLINICAL TRIAL: NCT01173575
Title: Assessment of the Efficacy of FOSFOMYCIN in Patients With Bacterial Infection
Status: Completed | Type: Observational
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: J&P Medical Research Ltd. (Other); Sandoz GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: J&P009SAN/2009
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2016-02

CONDITIONS: Bacterial Infection
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bacterial Infection: All Patients with bacterial infection receiving fosfomycin may be included

SUMMARY:
This project aims to assess the clinical and microbiological efficacy of fosfomycin(FOM) in patients with bacterial infection.

Primary objective:

• To assess clinical and microbiological efficacy of FOM in patients with bacterial infection.

Secondary objectives:

* To determine the rate and severity of unexpected adverse events.
* To determine the mean duration of therapy with FOM in patients with bacterial infection.

Study design:

Multi-center, non-interventional study

DETAILED DESCRIPTION:
Please note that InfectoPharm Arzneimittel und Consilium GmbH has taken over sponsor responsibilities for all German sites of this clinical trial with Jannuary 2016 from J&P MEDICAL RESEARCH LTD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bacterial infection receiving FOM for clinical purposes will be included into the analysis.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with bacterial infection considered suitable for routine antimicrobial therapy with FOM may be included into this analysis.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2010-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- Medical University Graz, Graz, Styria, Austria
- Germany (24):
  - University Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - Augsburg Hospital, Augsburg, Bavaria
  - Kreisklinik Guenzburg Krumbach, Krumbach, Bavaria
  - University Hospital Munich, Munich, Bavaria
  - University Hospital Regensburg, Regensburg, Bavaria
  - Weiden Hospital, Weiden in Der Oberpfalz, Bavaria
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Evangelische Krankenhausstiftung Oldenburg, Oldenburg, Lower Saxony
  - Klinikum Oldenburg gGmbH, Oldenburg, Lower Saxony
  - Klinikum Osnabrück, Osnabrück, Lower Saxony
  - University Hospital Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Heart and Diabetes Center North Rhine-Westphalia, Bad Oeynhausen, North Rhine-Westphalia
  - Medizinische Universitätsklinik Knappschaftskrankenhaus Bochum, Bochum, North Rhine-Westphalia
  - University of Bonn (Orthopedics), Bonn, North Rhine-Westphalia
  - University of Bonn (Anesthesiology), Bonn, North Rhine-Westphalia
  - University Hospital Cologne (Cardiothoracic Surgery), Cologne, North Rhine-Westphalia
  - University Hospital Cologne (Internal Medicine), Cologne, North Rhine-Westphalia
  - Hospital Cologne-Merheim, Cologne, North Rhine-Westphalia
  - University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Muenster, Münster, North Rhine-Westphalia
  - University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Vivantes Klinikum Neukölln, Berlin
  - Charite University Hospital Berlin, Berlin
  - Paulinenhaus Krankenanstalt e.V., Berlin

REFERENCES:
- [Derived] Putensen C, Ellger B, Sakka SG, Weyland A, Schmidt K, Zoller M, Weiler N, Kindgen-Milles D, Jaschinski U, Weile J, Lindau S, Kieninger M, Faltlhauser A, Jung N, Teschendorf P, Adamzik M, Grundling M, Wahlers T, Gerlach H, Litty FA. Current clinical use of intravenous fosfomycin in ICU patients in two European countries. Infection. 2019 Oct;47(5):827-836. doi: 10.1007/s15010-019-01323-4. Epub 2019 Jun 12. PMID 31190298